CLINICAL TRIAL: NCT00468234
Title: Validation of Biomarkers of Exposure and Host Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Institute for Science and Health (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 009-05
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cigarette Smoker
Keywords: smoking cessation; harm reduction; biomarker; exhaled breath condensate
MeSH Terms: conditions — Smoking Cessation; Harm Reduction | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Transdermal Patch; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: nicotine polacrilex
  Other Names: nicotine gum
Drug: nicotine transdermal system
  Other Names: patch
Drug: nicotine inhaler
  Other Names: nicotine oral inhaler

SUMMARY:
This study will evaluate biomarkers measured in exhaled breath condensate (EBC) to assess clinical strategies of harm reduction. It will take advantage of a recently developed device that permits collection of exhaled breath condensate reproducibly, with minimal subject effort and with no oral contamination. Samples from asymptomatic smokers before and after inducing a change in their smoking habit (cessation or reduction) with the aid of partial nicotine replacement.

DETAILED DESCRIPTION:
The proposed study will evaluate biomarkers measured in exhaled breath condensate (EBC) for the purpose of assessing clinical strategies of harm reduction. It will take advantage of a recently developed device that permits collection of exhaled breath condensate reproducibly, with minimal subject effort and with no oral contamination. The major goal of the trial is to provide evidence to validate biomarkers in EBC.

This will be accomplished by collecting samples from asymptomatic smokers before and after inducing a change in their smoking habit (cessation or reduction) with the aid of partial nicotine replacement.

Measures to be made in EBC include H2O2, the most widely explored biomarker in this "body" fluid. Methods that reliably can quantify levels in normal non-smokers and in asymptomatic smokers will be used. Two fold increases in smokers have been reported by in several reports and confirmed in preliminary data by the investigators. In addition, other biomarkers of oxidant stress: TBARs, 8-isoprostane and nitrotyrosine will be quantified using standard methods.

Biomarkers quantified in EBC will be assessed for reliability (i.e. reproducibility and for sensitivity) to change and for validity (by comparison to clinically defined endpoints and previously validated measures of exposure). Reproducibility will be assessed by making repeated measurements in the same subjects on different occasions. Sensitivity to change will be assessed by comparing values before and after changing smoking habit. Finally, the validity of the biomarkers will be assessed by comparing them to previous measures of smoke exposure (CO, NNAL and NNAL-glc) and to clinically defined endpoints: symptoms, the St. George's Respiratory Questionnaire and post bronchodilator lung function. With regard to the latter measures, preliminary data indicate that symptoms can be detected in "asymptomatic" smokers and that these can change with a harm reduction strategy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age or older
* Have a stable smoking habit greater than three months
* Have smoked for at least 5 pack years
* Be willing to make a serious quit attempt and be willing to use nicotine replacement therapy
* Be able to give informed consent

Exclusion Criteria:

* regular use of anti-inflammatory medication; presence of any inflammatory *disease of the respiratory tract including moderate or worse COPD (FEV1 < 80% predicted and FEV1/FVC ratio < 0.7) or PFT criteria for asthma (improvement in FEV1>12% of predicted and >200ml).
* Subjects with normal lung function who meet criteria for diagnosis of chronic bronchitis will be excluded.
* Subjects with stable medical conditions, excluding inflammatory lung disease, will be permitted to participate, providing anti-inflammatory therapies are not used regularly and providing there has been no change in their clinical status in the two months prior to beginning the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
exhaled breath hydrogen peroxide

SECONDARY OUTCOMES:
health status (SGRQ, CCQ, BCSS, LCQ)
lung function

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I Rennard, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States